CLINICAL TRIAL: NCT02893150
Title: Mindfulness as a Complementary Intervention for Overweight Primary Care Patients: Study Protocol for a Randomized Controlled Trial
Brief Title: Mindfulness Intervention for Overweight Primary Care Patients
Acronym: MindEat
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centro Mente Aberta de Mindfulness (Other)
Collaborators: Conselho Nacional de Desenvolvimento Científico e Tecnológico (Other Government)
Responsible Party: Principal Investigator, Marcelo Demarzo, MD, PhD, MD, Phd., Centro Mente Aberta de Mindfulness
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: Mindful Eating
Record Dates: First submitted 2016-08-29; First posted 2016-09-08 (Estimated); Last update posted 2021-10-15 (Actual); Status verified 2021-10

CONDITIONS: Overweight; Obesity
Keywords: Mindful Eating; Overweight; Primary Care; Randomized Clinical Trial
MeSH Terms: conditions — Overweight; Obesity

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- TAU (treatment as usual) (Active Comparator): The Treatment as Usual (TAU) will be considered as following: 1) In the cases of individuals presenting overweight (BMI of 25 kg/m ² to 29.9 kg/m ²), but without comorbidities, primary care teams propose the improvement of the life style (more physically active, and with a better eating behaviour) in order to return to the track of normal BMI (BMI of 18.5 kg/m ² to 24.9 kg/m ²). 2) For those who have comorbidities such as hypertension and diabetes, in addition to including individuals in group activities (psycho-education), it is evaluated the need for individual dietary prescription by a nutritionist.
  Interventions: Behavioral: TAU
- TAU+MBHP (Active Comparator): The Mindfulness-based Health Promotion (MBHP) developed by our research group (generic protocol) will be adapted from the Mindfulness-based Stress Reduction program (MBSR), It is based on the original model developed by Jon Kabat-Zinn and colleagues (MBSR), and subsequently adapted by our research group in order to fit it better into the context and needs of Primary Care (PC) and national and local Health Systems], which has been applied by the Center "Mente Aberta" in Brazil (www.mindfulnessbrasil.com), and by the University of Zaragoza, in Spain (www.webmindfulness.com). One of the sessions (the sixth one) is developed in silence, with the goal of deepening the mindfulness practice.
  Interventions: Behavioral: TAU+MBHP
- TAU+MB-EAT (Experimental): The Mindfulness-based Eating Awareness (MB-EAT) protocol consists in ten weekly sessions of 2,5 hour to improve compulsive eating, and to promote conscious eating.
  Interventions: Behavioral: TAU+MB-EAT

INTERVENTIONS:
Behavioral: TAU — TAU (Treatment as Usual), individuals presenting with overweight (BMI of 25 kg/m ² to 29.9 kg/m ²), but without comorbidities, teams of primary care (PC) organized care plans to return to the track of normal BMI (BMI of 18.5 kg/m ² to 24.9 kg/m ²).
  For those who have comorbidities such as hypertension and diabetes, in addition to including individuals in group activities, evaluates the need for individual dietary prescription by the nutritionist. This decision is discussed among the team of PC and Matrix support team
  Arms: TAU (treatment as usual)
Behavioral: TAU+MBHP — TAU (Treatment as Usual) + MBHP. We used a general (general vulnerability, not specific) mindfulness-based intervention (MBI) developed by our research group, an 8-week-group-based MBI called "Mindfulness-Based Health Promotion" (MBHP) program . It is based on the original model developed by Jon Kabat-Zinn and colleagues (MBSR), and subsequently adapted by our research group in order to fit it better into the context and needs of Primary Care (PC) and national and local Health Systems, which has been applied by the Center "Mente Aberta" in Brazil (www.mindfulnessbrasil.com), and by the University of Zaragoza, in Spain (www.webmindfulness.com). One of the sessions (the sixth one) is developed in silence, with the goal of deepening the mindfulness practice; more feasible to be implement in health services and facilities
  Arms: TAU+MBHP
Behavioral: TAU+MB-EAT — TAU (Treatment as Usual) + MB-EAT (mindfulness-based eating awareness training). Adapted from the MBSR, Mindfulness-based Eating Awareness Training (MB-EAT) or awareness training. This program was specially developed for the compulsive eating disorders and related problems[47]. In addition the four main techniques of meditation mentioned in the MBHP program includes modifications to these basic techniques, and include experimentation with different flavors, sweet and savory foods, etc. Has 10 weekly sessions of 2,5h
  Arms: TAU+MB-EAT

SUMMARY:
Mindfulness has been applied in the United States and Europe to improve both physical and psychological health, however, it is still poorly studied in Brazil. Mindfulness, or its lack, may also have particular relevance to obesity and eating disorders, reducing the episodes of "binge eating", which are partly responsible for weight regain for many people, and improving the eating behavior in order to promote awareness of emotional states which distort the physiological signals generated by the process. The hypothesis is that Mindfulness-based Interventions (MBI) as well as specific programmes focused on conscious eating, as Mindfulness Based Eating Awareness Training (MB-EAT) can, in short time, and in a sustainable fashion, improve biochemical, psychometric and anthropometric parameters in primary care patients with overweight.

DETAILED DESCRIPTION:
A randomized-controlled trial will be conducted to compare treatment-as-usual (TAU) in Primary Care combined a generic MBI (with 8 sessions) developed by our research group, called "Mindfulness-Based Health Promotion" (MBHP) program versus TAU plus MB-EAT. It will be included women aged ≥18 and < 60, literate , with a BMI (body mass index) ≥ 25 kg/m2. The primary outcome is the improvement of the eating behaviour measured by DEBQ. Secondary outcomes are: It is expected improvement of nutritional status (reduction of body weight by at least 5% of the weight) along the intervention, as well as maintenance of this (without weight regain) which could lead to the prevention of multiple morbidities related to excess body weight. Will be assessed the levels of Mindfulness, stress, anxiety (psychometric scale and serum cortisol) and self-compassion. There will be performed basal (baseline), at post-intervention, 3 and 6 months follow-up measurements. The control group will receive the intervention that has been shown to be more effective at the end of the study (MBHP or MB-EAT).

ELIGIBILITY:
Inclusion Criteria:

* women aged 18-59 years old, literate;
* Primary Care patients who have the body mass index (BMI) ≥25kgm2 and < 40kg/m2
* People who have an interest in the objectives of this study and consented to be randomized to one of three arms.
* Those who have participated in 75% of sessions or only two absences in the program

Exclusion Criteria:

* those who are under pharmacological treatment for overweight;
* pregnant women;
* those who have problems with substance use (drugs and alcohol);
* untreated hypothyroidism or hyperthyroidism;
* those who are in acute phase of depression (less than 6 months in depression); schizophrenia or psychotic disorders or who are using drugs that cause cognitive attentional and concentration losses (such as powerful anti-anxiety drugs);
* current practitioners of Mindfulness, meditation, yoga, or the like, in the last 6 months (with formal practice at least once a week);
* those who have undergone any type of Bariatric Surgery.

Ages: 18 Years to 59 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 284 (Actual)
Dates: Start 2018-04-05 (Actual); Primary Completion 2018-04-05 (Actual); Study Completion 2019-12-18 (Actual)

PRIMARY OUTCOMES:
Feeding Behaviour | Up to 3-month of follow-up
  It is expected the improvement of the feeding behaviour measured by Dutch Eating Behaviour Questionaire (DEBQ) in total score and in 3 subscales: Restriction , External Intake and Emotional Intake and with the scale EAT 26

SECONDARY OUTCOMES:
Fasting blood glucose | Up to 3-month of follow-up
  It is expected the improvement of Fasting blood glucose level
levels of mindfulness, | Up to 3-month of follow-up
  It expected to increase the levels of Mindfulness-psychometric scale
Levels of depression | Up to 3-month of follow-up
  It expected to reduce the levels of Depression-psychometric scale
Levels of anxiety | Up to 3-month of follow-up
  It expected to reduce the levels of anxiety -psychometric scale and serum cortisol
Serum cortisol | Up to 3-month of follow-up
  It expected to reduce the levels of cortisol
Self-compassion | Up to 3-month of follow-up
  It expected to improve the levels of self-compassion scale
HBA1C (glycated hemoglobina) | Up to 3-month of follow-up
  It is expected the improvement of glycated hemoglobina level
Insulin | Up to 3-month of follow-up
  It is expected reduction in insulin level

OTHER OUTCOMES:
Cholesterol and fractions, triglycerides | Up to 3-month of follow-up
  It is expected reduction in cholesterol and fractions level and triglycerides
C-reactive protein | Up to 3-month of follow-up
  It is expected reduction in PCR level
waist perimeter | Up to 3-month of follow-up
  It is expected reduction in waist perimeter
food consumption | Up to 3-month of follow-up
  It is expected improve quality of food consumption (questionaire)
Body fat | Up to 3-month of follow-up
  It is expected to reduce the body fat percentage (bioimpedance)
Basal metabolism rate | Up to 3-month of follow-up
  It is expected to increase the basal metabolic rate-calorimeter
Physical Activity | Up to 3-month of follow-up
  It is expected to increase the physical activity (Brief Physical Activity Assessment Tool
Risk of eating Disorder | Up to 3-month of follow-up
  It is expected to reduce the risk score of eating disorder (questionaire EAT 26)

CONTACTS AND LOCATIONS:
Overall Officials: Marcelo Demarzo, MD, PhD, Principal Investigator — UNIFESP - Federal University of Sao Paulo, Brazil
Locations (1):
- Centro Mente Aberta de Mindfulness e Promoção de Saúde, São Paulo, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Brasil. Ministério da Saúde. Secretaria de Atenção à Saúde. Departamento de Atenção Básica. Estratégias para o cuidado da pessoa com doença crônica : obesidade / Ministério da Saúde, Secretaria de Atenção à Saúde, Departamento de Atenção Básica. - Brasília : Ministério da Saúde, 2014. 212 p. : il. - (Cadernos de Atenção Básica, n. 38)- Academy of Nutrition and Dietetics. Weight Management Matters, 7 (4), Spring; 2010
- [Background] IBGE. Pesquisa de Orçamentos Familiares 2008-2009: análise do consumo alimentar pessoal no Brasil. Rio de Janeiro: Instituto Brasileiro de Geografia e Estatística, 2011
- [Background] Moura EC, Silva SA, Malta DC, Morais Neto OL. [Risk and protective factors for chronic non-communicable diseases: the VIGITEL telephone disease surveillance system, Brazil, 2007]. Cad Saude Publica. 2011 Mar;27(3):486-96. doi: 10.1590/s0102-311x2011000300009. Portuguese. PMID 21519699
- [Background] ______. Pesquisa de Orçamentos Familiares 2008-2009: análise do consumo alimentar pessoal no Brasil. Rio de Janeiro: Instituto Brasileiro de Geografia e Estatística, 2011.
- [Background] Prochaska JO, Velicer WF. The transtheoretical model of health behavior change. Am J Health Promot. 1997 Sep-Oct;12(1):38-48. doi: 10.4278/0890-1171-12.1.38. PMID 10170434
- [Background] Glanz K. Review of nutritional attitudes and counseling practices of primary care physicians. Am J Clin Nutr. 1997 Jun;65(6 Suppl):2016S-2019S. doi: 10.1093/ajcn/65.6.2016S. PMID 9174514
- [Background] De Nooijer J, Van Assema P, De Vet E, Brug J. How stable are stages of change for nutrition behaviors in the Netherlands? Health Promot Int. 2005 Mar;20(1):27-32. doi: 10.1093/heapro/dah504. Epub 2005 Jan 24. PMID 15668216
- [Background] Obesity: preventing and managing the global epidemic. Report of a WHO consultation. World Health Organ Tech Rep Ser. 2000;894:i-xii, 1-253. PMID 11234459
- [Background] Byrne S, Cooper Z, Fairburn C. Weight maintenance and relapse in obesity: a qualitative study. Int J Obes Relat Metab Disord. 2003 Aug;27(8):955-62. doi: 10.1038/sj.ijo.0802305. PMID 12861237
- [Background] Gusmão, J. L. et al. Adesão ao tratamento em hipertensão arterial sistólica isolada. Revista Brasileira de Hipertensão. 2009. 16(1): p. 38-43.
- [Background] Santos, A. C. A inserção do nutricionista na estratégia da saúde da família: o olhar de diferentes trabalhadores da saúde. Fam. Saúde Desenv. 2005.7(3): p.257-265.
- [Background] Oliveira DC, Sa CP, Gomes AM, Ramos Rde S, Pereira NA, Santos WC. [Brazilian National Health Policy: health professionals' social representations]. Cad Saude Publica. 2008 Jan;24(1):197-206. doi: 10.1590/s0102-311x2008000100020. Portuguese. PMID 18209848
- [Background] ______. Secretaria de Atenção à Saúde. Departamento de Atenção Básica. Política Nacional de Atenção Básica. Brasília: Ministério da Saúde, 2006f. (Série A. Normas e Manuais Técnicos), (Série Pactos pela Saúde, v. 4).
- [Background] Demarzo MMP. Mindfulness e Promoção da Saúde. RESC. 2015. 2(3): e82.
- [Background] Keng SL, Smoski MJ, Robins CJ. Effects of mindfulness on psychological health: a review of empirical studies. Clin Psychol Rev. 2011 Aug;31(6):1041-56. doi: 10.1016/j.cpr.2011.04.006. Epub 2011 May 13. PMID 21802619
- [Background] Camilleri GM, Mejean C, Bellisle F, Hercberg S, Peneau S. Association between Mindfulness and Weight Status in a General Population from the NutriNet-Sante Study. PLoS One. 2015 Jun 3;10(6):e0127447. doi: 10.1371/journal.pone.0127447. eCollection 2015. PMID 26038824
- [Background] Ludwig DS, Kabat-Zinn J. Mindfulness in medicine. JAMA. 2008 Sep 17;300(11):1350-2. doi: 10.1001/jama.300.11.1350. No abstract available. PMID 18799450
- [Background] Demarzo MMP. Meditação aplicada à saúde. Programa Atualização em Med Família e Comunidade. 6th ed. Porto Alegre-RS: Artmed. 2011. 6(1): p.1-18.
- [Background] Monshat K, Castle DJ. Mindfulness training: an adjunctive role in the management of chronic illness? Med J Aust. 2012 May 21;196(9):569-71. doi: 10.5694/mja11.10974. PMID 22621147
- [Background] Berg, Raquel. Uma análise freudiana da obesidade- Dissertação de Mestrado- programa de Pós-graduação em Psicologia da Universidade de São Paulo, 2008 136p.
- [Background] Brown KW, Ryan RM. The benefits of being present: mindfulness and its role in psychological well-being. J Pers Soc Psychol. 2003 Apr;84(4):822-48. doi: 10.1037/0022-3514.84.4.822. PMID 12703651
- [Background] Kaliman P, Alvarez-Lopez MJ, Cosin-Tomas M, Rosenkranz MA, Lutz A, Davidson RJ. Rapid changes in histone deacetylases and inflammatory gene expression in expert meditators. Psychoneuroendocrinology. 2014 Feb;40:96-107. doi: 10.1016/j.psyneuen.2013.11.004. Epub 2013 Nov 15. PMID 24485481
- [Background] Schutte NS, Malouff JM. A meta-analytic review of the effects of mindfulness meditation on telomerase activity. Psychoneuroendocrinology. 2014 Apr;42:45-8. doi: 10.1016/j.psyneuen.2013.12.017. Epub 2014 Jan 7. PMID 24636500
- [Background] Daubenmier J, Kristeller J, Hecht FM, Maninger N, Kuwata M, Jhaveri K, Lustig RH, Kemeny M, Karan L, Epel E. Mindfulness Intervention for Stress Eating to Reduce Cortisol and Abdominal Fat among Overweight and Obese Women: An Exploratory Randomized Controlled Study. J Obes. 2011;2011:651936. doi: 10.1155/2011/651936. Epub 2011 Oct 2. PMID 21977314
- [Background] Dalen J, Smith BW, Shelley BM, Sloan AL, Leahigh L, Begay D. Pilot study: Mindful Eating and Living (MEAL): weight, eating behavior, and psychological outcomes associated with a mindfulness-based intervention for people with obesity. Complement Ther Med. 2010 Dec;18(6):260-4. doi: 10.1016/j.ctim.2010.09.008. Epub 2010 Nov 11. PMID 21130363
- [Background] O'Reilly GA, Cook L, Spruijt-Metz D, Black DS. Mindfulness-based interventions for obesity-related eating behaviours: a literature review. Obes Rev. 2014 Jun;15(6):453-61. doi: 10.1111/obr.12156. Epub 2014 Mar 18. PMID 24636206
- [Background] Godfrey KM, Gallo LC, Afari N. Mindfulness-based interventions for binge eating: a systematic review and meta-analysis. J Behav Med. 2015 Apr;38(2):348-62. doi: 10.1007/s10865-014-9610-5. Epub 2014 Nov 23. PMID 25417199
- [Background] Satter E. Eating competence: definition and evidence for the Satter Eating Competence model. J Nutr Educ Behav. 2007 Sep-Oct;39(5 Suppl):S142-53. doi: 10.1016/j.jneb.2007.01.006. PMID 17826695
- [Background] Mantzios M, Wilson JC. Mindfulness, Eating Behaviours, and Obesity: A Review and Reflection on Current Findings. Curr Obes Rep. 2015 Mar;4(1):141-6. doi: 10.1007/s13679-014-0131-x. PMID 26627097
- [Background] Olson KL, Emery CF. Mindfulness and weight loss: a systematic review. Psychosom Med. 2015 Jan;77(1):59-67. doi: 10.1097/PSY.0000000000000127. PMID 25490697
- [Background] Katterman SN, Kleinman BM, Hood MM, Nackers LM, Corsica JA. Mindfulness meditation as an intervention for binge eating, emotional eating, and weight loss: a systematic review. Eat Behav. 2014 Apr;15(2):197-204. doi: 10.1016/j.eatbeh.2014.01.005. Epub 2014 Feb 1. PMID 24854804
- [Background] Academy of Nutrition and Dietetics. Weight Management Matters, 7 (4), Spring; 2010
- [Background] Kristeller JL, Wolever RQ. Mindfulness-based eating awareness training for treating binge eating disorder: the conceptual foundation. Eat Disord. 2011 Jan-Feb;19(1):49-61. doi: 10.1080/10640266.2011.533605. PMID 21181579
- [Background] Kristeller, J. L. Mindfulness, wisdom and eating: Applying a multi-domain model of meditation effects. Journal of Constructivism in the Human Sciences, 2003. 8: p. 107-118.
- [Background] Black DS, Semple RJ, Pokhrel P, Grenard JL. Component Processes of Executive Function-Mindfulness, Self-control, and Working Memory-and Their Relationships with Mental and Behavioral Health. Mindfulness (N Y). 2011 Sep;2(3):179-185. doi: 10.1007/s12671-011-0057-2. PMID 22013495
- [Background] Hill CL, Updegraff JA. Mindfulness and its relationship to emotional regulation. Emotion. 2012 Feb;12(1):81-90. doi: 10.1037/a0026355. Epub 2011 Dec 12. PMID 22148996
- [Background] Chiesa A, Malinowski P. Mindfulness-based approaches: are they all the same? J Clin Psychol. 2011 Apr;67(4):404-24. doi: 10.1002/jclp.20776. Epub 2011 Jan 19. PMID 21254062
- [Background] Goyal M, Singh S, Sibinga EM, Gould NF, Rowland-Seymour A, Sharma R, Berger Z, Sleicher D, Maron DD, Shihab HM, Ranasinghe PD, Linn S, Saha S, Bass EB, Haythornthwaite JA. Meditation programs for psychological stress and well-being: a systematic review and meta-analysis. JAMA Intern Med. 2014 Mar;174(3):357-68. doi: 10.1001/jamainternmed.2013.13018. PMID 24395196
- [Background] Green, S. M., & Bieling, P. J. Expanding the scope of mindfulness-based cognitive therapy: Evidence for effectiveness in a heterogeneous psychiatric sample. Cognitive and Behavioral Practice, 2012. 19(1): p.174- 180.
- [Background] Hofmann SG, Sawyer AT, Witt AA, Oh D. The effect of mindfulness-based therapy on anxiety and depression: A meta-analytic review. J Consult Clin Psychol. 2010 Apr;78(2):169-83. doi: 10.1037/a0018555. PMID 20350028
- [Background] Alberts HJ, Mulkens S, Smeets M, Thewissen R. Coping with food cravings. Investigating the potential of a mindfulness-based intervention. Appetite. 2010 Aug;55(1):160-3. doi: 10.1016/j.appet.2010.05.044. Epub 2010 May 21. PMID 20493913
- [Background] Caldwell K, Baime M, Wolever R. Mindfulness based approaches to obesity and weight loss maintenance. J Men Health Couns, 2012. 34: p.269.
- [Background] Niemeier HM, Leahey T, Palm Reed K, Brown RA, Wing RR. An acceptance-based behavioral intervention for weight loss: a pilot study. Behav Ther. 2012 Jun;43(2):427-35. doi: 10.1016/j.beth.2011.10.005. Epub 2011 Dec 1. PMID 22440077
- [Background] Forman EM, Butryn ML, Juarascio AS, Bradley LE, Lowe MR, Herbert JD, Shaw JA. The mind your health project: a randomized controlled trial of an innovative behavioral treatment for obesity. Obesity (Silver Spring). 2013 Jun;21(6):1119-26. doi: 10.1002/oby.20169. Epub 2013 May 13. PMID 23666772
- [Background] Moher D, Hopewell S, Schulz KF, Montori V, Gotzsche PC, Devereaux PJ, Elbourne D, Egger M, Altman DG. CONSORT 2010 explanation and elaboration: updated guidelines for reporting parallel group randomised trials. BMJ. 2010 Mar 23;340:c869. doi: 10.1136/bmj.c869. No abstract available. PMID 20332511
- [Background] Zwarenstein M, Treweek S, Gagnier JJ, Altman DG, Tunis S, Haynes B, Oxman AD, Moher D; CONSORT group; Pragmatic Trials in Healthcare (Practihc) group. Improving the reporting of pragmatic trials: an extension of the CONSORT statement. BMJ. 2008 Nov 11;337:a2390. doi: 10.1136/bmj.a2390. PMID 19001484
- [Background] Cordás TA, Neves JEP. Escalas de avaliação de transtornos alimentares. Rev Psiq Clin. 1999, 26: p. 41-8.
- [Background] Cordás TA, Hochgraf PO. "BITE": instrumento para avaliação da bulimia nervosa - versão português. J Bras Psiquiatr ,1993. 42: p.141-4.
- [Background] Castro M, Moreira AC. Análise Crítica do Cortisol Salivar na Avaliação do Eixo Hipotálamo-Hipófise-Adrenal. Arq Bras Endocrinol Metab, 2003.7(4):p. 358-367.
- [Background] Raff H. Salivary cortisol: a useful measurement in the diagnosis of Cushing's syndrome and the evaluation of the hypothalamic-pituitary-adrenal axis. The Endocrinologist, 2000. 10: p. 9-17.
- [Background] de Salvo VL, Gimeno SG. [Reproducibility and validity of a food frequency questionnaire]. Rev Saude Publica. 2002 Aug;36(4):505-12. doi: 10.1590/s0034-89102002000400018. Portuguese. PMID 12364926
- [Background] Duarte, A. C. et al. Síndrome metabólica: semiologia, bioquímica e prescrição nutricional. Rio de Janeiro: Axcel Books do Brasil, 2005.
- [Background] Faria SL, Faria OP, Cardeal MD, Ito MK. Validation study of multi-frequency bioelectrical impedance with dual-energy X-ray absorptiometry among obese patients. Obes Surg. 2014 Sep;24(9):1476-80. doi: 10.1007/s11695-014-1190-5. PMID 24464546
- [Background] Rodrigues AE, Marostegan PF, Mancini MC, Dalcanale L, Melo ME, Cercato C, Halpern A. [Analysis of resting metabolic rate evaluated by indirect calorimetry in obese women with low and high caloric intake]. Arq Bras Endocrinol Metabol. 2008 Feb;52(1):76-84. doi: 10.1590/s0004-27302008000100011. Portuguese. PMID 18345399
- [Background] Melo CM, Tirapegui J, Ribeiro SM. [Human energetic expenditure: concepts, assessment methods and relationship to obesity]. Arq Bras Endocrinol Metabol. 2008 Apr;52(3):452-64. doi: 10.1590/s0004-27302008000300005. Portuguese. PMID 18506270
- [Background] Barros, V. V., E. H. Kozasa, I. C. W. Souza and T. M. Ronzani .
- [Background] Neff, K. The development and validation of a scale to measure self-compassion. Self and Identity, 2003a. 2: p. 85-101.
- [Background] Neff, K. Self-Compassion: An Alternative Conceptualization of a Healthy Attitude Toward Oneself. Self and Identity, 2003. 2: p. 85-101.
- [Background] Neff, K. Self-compassion and adaptive psychological functioning. Journal of Research in Personality, 2007. 41: p. 139-154.
- [Background] Neff KD, Germer CK. A pilot study and randomized controlled trial of the mindful self-compassion program. J Clin Psychol. 2013 Jan;69(1):28-44. doi: 10.1002/jclp.21923. Epub 2012 Oct 15. PMID 23070875
- [Background] BECK AT, WARD CH, MENDELSON M, MOCK J, ERBAUGH J. An inventory for measuring depression. Arch Gen Psychiatry. 1961 Jun;4:561-71. doi: 10.1001/archpsyc.1961.01710120031004. No abstract available. PMID 13688369
- [Background] Cunha, J. A. Manual da versão em português das Escalas Beck. São Paulo: Casa do Psicólogo, 2001.
- [Background] Queiroz DT, Vall J, Souza AMA, Vieira NFC. Observação participante na pesquisa qualitativa: conceitos e aplicações na área da saúde. R Enferm UERJ, 2007.15(2): p.276-83.
- [Background] Kerrigan D, Johnson K, Stewart M, Magyari T, Hutton N, Ellen JM, Sibinga EM. Perceptions, experiences, and shifts in perspective occurring among urban youth participating in a mindfulness-based stress reduction program. Complement Ther Clin Pract. 2011 May;17(2):96-101. doi: 10.1016/j.ctcp.2010.08.003. Epub 2010 Sep 16. PMID 21457899
- [Background] Nakamura E. O Método Etnográfico em Pesquisas na Área da Saúde: uma reflexão antropológica Saúde Soc. São Paulo, 2011. 20(1): p.95-103.
- [Result] Sociedade Brasileira de Endocrinologia e Metabologia- Projeto Diretrizes - Obesidade: Terapia Cognitivo-Comportamental, 2005 10p.
- [Derived] Salvo V, Schveitzer MC, Sanudo A, Favarato ML, Demarzo M. Exploring perceptions about Mindfulness and Mindful Eating Programs for low-income women with overweight in primary health care. Nutr Health. 2023 Jun;29(2):319-329. doi: 10.1177/02601060221075537. Epub 2022 Feb 9. PMID 35138182
- [Derived] Salvo V, Kristeller J, Montero Marin J, Sanudo A, Lourenco BH, Schveitzer MC, D'Almeida V, Morillo H, Gimeno SGA, Garcia-Campayo J, Demarzo M. Mindfulness as a complementary intervention in the treatment of overweight and obesity in primary health care: study protocol for a randomised controlled trial. Trials. 2018 May 11;19(1):277. doi: 10.1186/s13063-018-2639-y. PMID 29751819